CLINICAL TRIAL: NCT05920226
Title: Myocardial Fibrosis in Patients With Permanent Pacemakers
Status: Active, not recruiting | Type: Observational
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Principal Investigator, Suchkov Igor A., Professor, Ryazan State Medical University
Other Study IDs: Fibrosis05/23
Record Dates: First submitted 2023-06-13; First posted 2023-06-27 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Fibrosis; Atrial Fibrillation; Atrial Flutter
MeSH Terms: conditions — Fibrosis; Atrial Fibrillation; Atrial Flutter | interventions — Electrocardiography; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Extraction of peripheral venous blood to determine the level of myocardial fibrosis markers (Halitin-3, ST2);
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- A: 150 patients with indications for pacemakers implantation;: * men or women over 60 years of age
  * with signed informed consent form
  * in presence of cardiac pathology and arrhythmia requiring pacemakers implantation.
  * without active cancer or remission period less than 5 years;
  * without decompensated somatic pathology;
  * without active viral hepatitis, HIV or syphilis.
  Patients will be under observation for 2 years (inclusion in the study, visit 1, 12, 24 months after inclusion in the study).
  Interventions: Device: pacemakers implantation and assessment of cardiac function and cardiac fibrosis
- B: 150 patients without pacemakers implantation;: * men or women over 60 years of age
  * with signed informed consent form
  * in presence of cardiac pathology and arrhythmia not requiring pacemaker implantation.
  * without active cancer or remission period less than 5 years;
  * without decompensated somatic pathology;
  * without active viral hepatitis, HIV or syphilis.
  Interventions: Diagnostic Test: assessment of cardiac function and cardiac fibrosis

INTERVENTIONS:
Device: pacemakers implantation and assessment of cardiac function and cardiac fibrosis — 150 patients will be implanted with pacemakers. In addition to the echocardiography, contrast-enhanced cardiac MRI and peripheral venous blood sampling for myocardial fibrosis markers, the tests described above will be repeated at 1 (V1), 12 (V2), 24 (V3) months after inclusion. Echocardiography and peripheral venous blood sampling for myocardial fibrosis markers detection will be repeated to all patients before pacemakers implantation and after 6,12 and 24 months of observation period. Contrast-enhanced cardiac magnetic resonance imaging (MRI) will be performed before pacemaker implantation and 6 months after surgery.
  In addition, pacemakers programming data will be evaluated after 1, 12, 24 months after inclusion in the study (atrioventricular delay, percentage of ventricular stimulation, episodes of high atrial frequency, fibrillation/atrial flutter, ventricular tachycardia).
  Other Names: Withdrawal of Peripheral venous blood samples; electrocardiography; echocardiography; contrast-enhanced cardiac MRI
  Groups: A: 150 patients with indications for pacemakers implantation;
Diagnostic Test: assessment of cardiac function and cardiac fibrosis — The patients who do not require a pacemaker placement will undergo diagnostic testing such as echocardiography, contrast-enhanced cardiac MRI and peripheral venous blood sampling for myocardial fibrosis markers.
  Other Names: Withdrawal of Peripheral venous blood samples; electrocardiography; echocardiography; contrast-enhanced cardiac MRI
  Groups: B: 150 patients without pacemakers implantation;

SUMMARY:
Patients with cardiac pathology and arrhythmias including those who have indications for pacemakers implantation will be included in the study. We will determine the influence of pacemaker implantation with the localization of the ventricular electrode in the top of the right ventricle or the middle third of the right ventricle according to echocardiographic and electrocardiographic parameters, congestive heart failure progression, patients' quality of life and follow-up therapy of patients with identified myocardial fibrosis with existing pacemaker.

Study of changes in echocardiography, electrocardiography, myocardial fibrosis markers, the quality of life of patients will allow to choose the most optimal localization of the ventricular electrode during implantation of the permanent pacemakers system in order to improve the quality of life of the patients.

DETAILED DESCRIPTION:
Anticipated design of the study: an open, prospective, study, with parallel groups of patients according to ICH GCP ((International Conference on Harmonisation - Good Clinical Practice) criteria.

The study will involve 300 patients with cardiac pathology and arrhythmias including those who have indications for pacemakers implantation, who will be allocated into 2 groups: group 1 - patients who require a permanent pacemaker placement; group 2 - patients who do not require a permanent pacemaker placement.

Patients involved in the study will undergo peripheral venous blood sampling to determine the level of myocardial fibrosis markers (Halitin-3, ST2), electrocardiography (assessment of the type of bradyarrhythmia, assessment of the presence/absence and type of intraventricular conductivity disorder, estimation of the width of the QRS complex, direction of the electric axis of the heart), echocardiography (evaluation of ejection fraction, heart chamber size, mitral and tricuspidal manifestation, interventricular delay), contrast-enhanced cardiac magnetic resonance imaging (MRI), quality of life assessment using the Aquarel questionnaire. All procedures will be repeated at time points as per protocol.

Specific information for Group A patients: there will be different variants of localization of the right ventricular lead (top of the right ventricle, the upper third of the ventricular septum, the middle third of the ventricular septum, the lower third of the ventricular septum, front wall of the right ventricle, lower wall of the right ventricle, parahisial region, His bundle). The analysis of the subgroups will be carried out according to the following criteria: electrode localization, main indication for pacemakers implantation, pacemakers model, type of initial intraventricular conductivity disorder.

ELIGIBILITY:
Inclusion Criteria:

1. men or women over 60 years of age
2. . signed informed consent form
3. . presence of cardiac pathology and arrhythmia requiring pacemakers implantation (group A).
4. . presence of cardiac pathology and arrhythmia not requiring pacemaker implantation (group B).

Exclusion Criteria:

1. . active cancer or remission period less than 5 years;
2. . decompensated somatic pathology;
3. . active viral hepatitis, HIV or syphilis;
4. . men or women younger than 60 years of age or older than 85 years of age;
5. . withdrawn consent.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 150 patients with cardiac pathology and arrhythmia not requiring pacemaker implantation and 150 patients with cardiac pathology and arrhythmia requiring pacemaker implantation (with different localization of the right ventricular lead).
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes in indicators of myocardial fibrosis | June 2023 - June 2028
  Changes in indicators of myocardial fibrosis in patients with cardiac arrhythmias depending on type of treatment

SECONDARY OUTCOMES:
Changes in echocardiography parameters | June 2023 - June 2028
  Changes in echocardiography parameters such as ejection fraction, valve regurgitation.
Changes in quality of life | June 2023 - June 2028
  Changes in quality of life in patients with cardiac arrhythmias depending on type of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Igor Suchkov, MD DMedSc, Principal Investigator — Ryazan State Medical University
Locations (1):
- Ryazan State Medical University, Ryazan, Russia